CLINICAL TRIAL: NCT05438537
Title: A Comprehensive Prospective Assessment of the Physical and Biological Effects of Upper Tract Urothelial Cancer (UTUC)
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2020.484
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Upper Tract Urothelial Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are many controversies and limitations in the management of Upper Tract Urothelial cancer. A prospective registry is set up for patients in our hospital, aim to have a comprehensive prospective assessment of the physical and biological effects of Upper Tract Urothelial cancer in our patients

DETAILED DESCRIPTION:
Although Upper Tract Urothelial Carcinoma (UTUC) is relatively uncommon, the incidence rate is increasing. There are many controversies and limitations in the management of Upper Tract Urothelial cancer.

In this study, investigators would like to establish a local registry for upper tract urothelial cancer to facilitate the collection of clinical information and outcomes of upper tract urothelial cancer management, and to collect blood, urine and tumour tissue samples to investigate for new diagnostic and therapeutic agents. Hopefully, our registry can provide information regarding the epidemiology, natural history, and treatment outcomes of upper tract urothelial cancer in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Male patients > 18 years old
* Patients who has presence of UTUC and pending for surgery
* Patients who has history of UTUC with any intervention performed

Exclusion Criteria:

- Patients fail to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 300 Chinese patients with various stage of UTUC will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Long-term survival | 10 years
  Long-term survival

SECONDARY OUTCOMES:
Recurrence rate of UTUC | 10 years
  Recurrence rate of UTUC
Progression rate of UTUC | 10 years
  Progression rate of UTUC
Complications | 10 years
  Complications are assessed by medical record and on patient follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Yuen-Chun TEOH, FRCS(Ed) MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cauberg EC, Salomons MA, Kummerlin IP, de Reijke TM, Zwinderman AH, de la Rosette JJ, Kate FJ, Laguna Pes MP. Trends in epidemiology and treatment of upper urinary tract tumours in the Netherlands 1995-2005: an analysis of PALGA, the Dutch national histopathology registry. BJU Int. 2010 Apr;105(7):922-7. doi: 10.1111/j.1464-410X.2009.08889.x. Epub 2009 Oct 5. PMID 19804428
- [Background] Lughezzani G, Burger M, Margulis V, Matin SF, Novara G, Roupret M, Shariat SF, Wood CG, Zigeuner R. Prognostic factors in upper urinary tract urothelial carcinomas: a comprehensive review of the current literature. Eur Urol. 2012 Jul;62(1):100-14. doi: 10.1016/j.eururo.2012.02.030. Epub 2012 Feb 23. PMID 22381168
- [Background] Mellemgaard A, Carstensen B, Norgaard N, Knudsen JB, Olsen JH. Trends in the incidence of cancer of the kidney, pelvis, ureter and bladder in Denmark 1943-88. Scand J Urol Nephrol. 1993;27(3):327-32. doi: 10.3109/00365599309180442. PMID 8290911
- [Background] Munoz JJ, Ellison LM. Upper tract urothelial neoplasms: incidence and survival during the last 2 decades. J Urol. 2000 Nov;164(5):1523-5. PMID 11025695
- [Background] Remzi M, Shariat S, Huebner W, Fajkovic H, Seitz C. Upper urinary tract urothelial carcinoma: what have we learned in the last 4 years? Ther Adv Urol. 2011 Apr;3(2):69-80. doi: 10.1177/1756287211403349. PMID 21869907